CLINICAL TRIAL: NCT01582893
Title: Permeability Enhancement to Reduce Chronic Inflammation
Acronym: PERCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1492; CIV-11-10-002741 (Other: Eudamed)
Record Dates: First submitted 2012-04-11; First posted 2012-04-23 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Inflammation
Keywords: inflammation; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCO1100-P14L (Experimental): HCO1100 is connected in row with low flux dialyzer P14L
  Interventions: Device: HCO1100
- P210H (Active Comparator): High flux Filter P210H
  Interventions: Device: P210H

INTERVENTIONS:
Device: HCO1100 — Dialysis
  Arms: HCO1100-P14L
Device: P210H — Dialysis
  Arms: P210H

SUMMARY:
Chronic dialysis patients with end stage renal disease have an increased mortality rate as compared to the age matched healthy population. It is known that chronic inflammation contributes to the high incidence of cardiovascular events in chronic dialysis patients. Dialyzers made by membranes with increased pore size (high cut-off Dialyzer HCO1100) may be beneficial in the elimination of inflammatory mediators and may improve the inflammatory status. Hypothesis: In this study it will be investigated whether the treatment with HCO1100 will improve the inflammatory status of chronic dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis treatment for ≥ 3 months
* Dialysis 3x weekly
* Vascular access by fistula or CVC providing QB of ≥ 250 ml/min
* Dialysis with high-flux dialyzer for a minimum of 2 weeks before begin of study
* CRP > 5mg/L at least once within 12 weeks before inclusion
* Age > 18 and < 99 Years
* Ability to give written informed consent

Exclusion Criteria:

* Missing informed consent form
* Clinically manifested infection or current CRP-value > 50mg/L
* Serum albumin < 35g/L
* Intake of immune suppressive medication
* Pregnancy or lactation
* Participation in a different study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change of CD162 expression on monocytes | 8 weeks (3 weeks treatment phase, 2 weeks wash out phase, 3 weeks treatment phase)
  change of CD162 expression on monocytes, timepoints in each treatment phase: 1.)1st.day (prae dialysis) 2.)1st.day (post dialysis) 3.)2nd.day (prae dialysis) 4.)8th.day (prae dialysis) 5.)15th.day (prae dialysis) 6.)22nd.day (prae dialysis)

SECONDARY OUTCOMES:
Albumin blood level | 8 weeks (3 weeks treatment phase, 2 weeks wash out phase, 3 weeks treatment phase)
  change of albumin blood level, timepoints in each treatment phase: 1.)1st.day (prae dialysis) 2.)1st.day (post dialysis) 3.)2nd.day (prae dialysis) 4.)8th.day (prae dialysis) 5.)15th.day (prae dialysis) 6.)22nd.day (prae dialysis)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Girndt, MD, Study Director — Martin-Luther-Universität Halle-Wittenberg; Ralf Schindler, MD, Principal Investigator — Charité, Humboldt Universität Berlin
Locations (2):
- Germany (2):
  - KfH Bachstzelzenweg 4, Halle, Saxony-Anhalt
  - KfH-Bismarkstrasse 95-96, Berlin